CLINICAL TRIAL: NCT03007914
Title: A Multi-center, Prospective, Cohort Study to Evaluate the Effectiveness of Traditional Chinese Medicine on COPD Patients
Brief Title: Effect of Traditional Chinese Medicine on Outcomes in COPD Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Henan University of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: TCM for COPD Cohort
Record Dates: First submitted 2016-12-26; First posted 2017-01-02 (Estimated); Last update posted 2017-01-02 (Estimated); Status verified 2016-12

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Pulmonary Disease, Chronic Obstructive; Medicine, Chinese Traditional; Humans; Treatment Outcome
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — The biological sample bank includes serum samples, plasma samples, sputum samples, urine samples, stool samples.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- TCM cohort: Patients continue to receive the routine TCM treatments recommended by 2011 Chinese treatment guidelines of TCM for COPD.
- Conventional medicine cohort: Patients continue to receive the conventional medicine recommended by 2014 GOLD and Chinese treatment guidelines for COPD.

SUMMARY:
The aim of this study is to compare the effectiveness of the treatments in two cohort for COPD patients: one, traditional Chinese medicine (TCM) cohort, which have been evaluated and have certain effect; the other, conventional medicine treatments cohort, based on 2015 Global Initiative for Chronic Obstructive Lung Disease (GOLD).

DETAILED DESCRIPTION:
COPD, with high prevalence, morbidity, mortality and economic burdens, affects millions worldwide. Although many therapies exist and are being developed to relieve symptoms and reduce mortality in COPD, most have only been studied in placebo-controlled efficacy studies in highly selected populations. There are few clinical trials to compare therapeutic alternatives in real world. Furthermore, some randomized controlled trials on comprehensive TCM interventions, especially based on the TCM patterns, have been the certain evidence for showing definite effect for COPD patients. In addition, studies in real world populations of COPD that received different therapies that do have efficacy evidence was found wide variations in care delivery. In short, there is a need for cohort study in COPD.

This is a multi-center, prospective, cohort study to evaluate the effectiveness of TCM on COPD patients. The cohort study will enroll approximately 2540 patients that in two cohort, one, TCM cohort, which have been evaluated and have certain effect; the other, conventional medicine treatments cohort, based on 2015 Global Initiative for Chronic Obstructive Lung Disease (GOLD).Subjects in two cohort will be followed-up 2 years.The primary outcome measure is the frequency of exacerbations. The secondary efficacy measures include mortality rate and all-cause mortality, FEV1, dyspnea (MMRC), exercise capacity( 6MWD), quality of life ( CAT, SF-36 and COPD-PRO), and effectiveness satisfaction with treatment(ESQ-COPD).

ELIGIBILITY:
Inclusion Criteria:

* A confirmed diagnosis of COPD.
* Medically stable.
* Age between 40 and 80 years.
* Syndrome differentiation belongs to syndrome of deficiency of deficiency of lung qi, deficiency of pulmonic-splenic qi, syndrome of insufficiency of qi of the lung and kidney, syndrome of insufficiency of qi and yin of the lung and kidney.
* With the informed consent signed.
* Capable of complying with the dosing regimen and visit schedules.

Exclusion Criteria:

* Pregnant or breast-feeding women.
* Any psychiatric condition rendering the patient unable to understand the nature, scope and possible consequences of the study.
* Malignancy for which patient has undergone resection, radiation therapy or chemotherapy within the last 5 years.
* Current respiratory disorders other than COPD (e.g., bronchiectasis, bronchial asthma, tuberculosis, lung fibrosis, pulmonary thromboembolic, diffuse panbronchiolitis).
* Complicated with heart failure (NYHA Class III or IV),or myocardial infarction within six months ,or unstable hemodynamics.
* Complicated with serious hepatic and renal diseases (liver cirrhosis, portal hypertension, bleeding of varicose veins, dialysis, or renal transplantation).
* Complicated with congenital or acquired immune deficiency.
* Participating in other trials or allergic to the used medicine.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: COPD patients
Sampling Method: Probability Sample
Enrollment: 2540 (Estimated)
Dates: Start 2016-12; Primary Completion 2020-05 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
The frequency of exacerbation | Change from Baseline in the frequency of exacerbation at the months 3, 6, 9, 12, 15, 18, 21, and 24 of the follow up phase.

SECONDARY OUTCOMES:
All cause mortality | The all-cause mortality in 2 years of the follow up phase.
Forced expiratory volume in one second | Change from Baseline in the one second (FEV1) at the months 3, 6, 9, 12, 15, 18, 21, and 24 of the follow up phase.
  FEV1 is the amount of air that can be exhaled in one second.
Dyspnea | Change from Baseline in MMRC at the months 3, 6, 9, 12, 15, 18, 21, and 24 of the follow up phase.
  Using Modified Medical Research Council (MMRC) scale to assess a patient's level of dyspnea. The MMRC scale is a simple grading system that scored from 0 (less severe) to 4 (severe).
Minutes Walking Distance Test (6MWD) | Change from Baseline in the 6MWD at the months 3, 6, 9, 12, 15, 18, 21, and 24 of the follow up phase.
COPD Assessment Test (CAT) | Change from Baseline in the CAT at the months 3, 6, 9, 12, 15, 18, 21, and 24 of the follow up phase.
  Using the CAT to evaluate the impact of COPD on a person's life over time.
Effectiveness satisfaction with treatment | Change from Baseline in the ESQ-COPD at the months 3, 6, 9, 12, 15, 18, 21, and 24 of the follow up phase.
  Using the effectiveness satisfaction questionnaire of chronic obstructive pulmonary disease (ESQ-COPD) to evaluate COPD patients' satisfaction with their treatment over time.
Short Form 36-Item Health Survey (SF-36) | Change from Baseline in the SF-36 at the months 3, 6, 9, 12, 15, 18, 21, and 24 of the follow up phase.
  Using the SF-36 to evaluate the impact of COPD on a person's life over time.
Patient reported outcome for COPD (COPD-PRO) | Change from Baseline in the COPD-PRO at the months 3, 6, 9, 12, 15, 18, 21, and 24 of the follow up phase.
  Using the COPD-PRO to evaluate the impact of COPD on a person's life over time.

CONTACTS AND LOCATIONS:
Overall Officials: Jiansheng Li, Doctor, Study Chair — The First Affiliated Hospital of Henan University of Traditional Chinese Medicine

IPD SHARING:
Plan to Share IPD: No